CLINICAL TRIAL: NCT06728592
Title: Emergency Stroke Unit for Acute Cerebrovascular Events: A Prospective, Single-arm Trial With a Historical Control Group
Acronym: ESU-ACE-E
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Leung Wai Hong Thomas, Professor, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Crec No. 2024.400T
Record Dates: First submitted 2024-12-05; First posted 2024-12-11 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Ischemic Stroke; Intracerebral Hemorrhage; Stroke; Stroke, Acute; Stroke, Ischemic; Stroke Hemorrhagic; Stroke (CVA) or TIA; Brain Diseases
MeSH Terms: conditions — Ischemic Stroke; Cerebral Hemorrhage; Stroke; Hemorrhagic Stroke; Brain Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Acute ischemic stroke patients , potentially eligible for IVT and/or EVT (Experimental): Acute ischemic stroke patients who are potentially eligible for IVT and/or EVT therapies and can be treated within 6 hours of symptom onset, will be triaged for intravenous thrombolysis (IVT) and/or endovascular thrombectomy (EVT) in Emergency Stroke Unit (ESU) based on lfMRI for diagnosis of ischemic stroke, differentiation of intracerebral hemorrhage (ICH) and identification of large vessel occlusion (LVO). Other screening and assessment procedures for IVT/EVT, and clinical management of the patients, are the same with standard practice as recommended by contemporary guidelines. In the historical control group, patients were triaged for IVT and/or EVT by standard practice, using plain CT and CTA for imaging triage.
  Interventions: Device: Portable Magnetic Resonance Imaging

INTERVENTIONS:
Device: Portable Magnetic Resonance Imaging — 0.23T Low-field Magnetic Resonance Imaging
  Other Names: Low-field Magnetic Resonance Imaging

SUMMARY:
Background Reperfusion therapies, i.e., intravenous thrombolysis (IVT) and/or endovascular thrombectomy (EVT), are most effective treatments in the management of acute ischemic stroke (AIS) patients. The benefits of reperfusion therapies, however, may be reduced by treatment delays due to tests and examinations and logistic issues. Emergency Stroke Unit (ESU), a new concept of stroke unit locating at the Accident and Emergency Department (AED), equipped with a mobile, low-field MR imaging (lfMRI) scanner for fast diagnosis of ischemic stroke, differentiation of intracranial hemorrhage and identification of large vessel occlusion (LVO), is being tested in Mainland China. It may shorten the door-to-needle time (DNT) for IVT and door-to-groin puncture time (DPT) for EVT, which may hance associate with improved functional outcomes of AIS patients.

This is a prospective, single-center, open-label, non-randomized, single-arm study aims to evaluate the safety and efficacy of the ESU workflow using lfMRI in shortening the DNT/DPT and improving functional outcomes in AIS patients, who are potentially eligible for IVT and/or EVT and can be treated within 6 hours after onset, compared with standard practice in Hong Kong; to reveal the changes in the ischemic lesions over a few days after IVT/EVT in these patients, with serial follow-up lfMRI exams.

DETAILED DESCRIPTION:
Background:

Reperfusion therapies, i.e., intravenous thrombolysis (IVT) and/or endovascular thrombectomy (EVT), are most effective treatments in the management of acute ischemic stroke (AIS) patients. The benefits of reperfusion therapies, however, may be reduced by treatment delays due to tests and examinations and logistic issues. Emergency Stroke Unit (ESU), a new concept of stroke unit locating at the Accident and Emergency Department (AED), equipped with a mobile, low-field MR imaging (lfMRI) scanner for fast diagnosis of ischemic stroke, differentiation of intracranial hemorrhage and identification of large vessel occlusion (LVO), is being tested in Mainland China. It may shorten the door-to-needle time (DNT) for IVT and door-to-groin puncture time (DPT) for EVT, which may hance associate with improved functional outcomes of AIS patients.

Objectives:

To evaluate the safety and efficacy of the ESU workflow using lfMRI in shortening the DNT/DPT and improving functional outcomes in AIS patients, who are potentially eligible for IVT and/or EVT and can be treated within 6 hours after onset, compared with standard practice in Hong Kong; to reveal the changes in the ischemic lesions over a few days after IVT/EVT in these patients, with serial follow-up lfMRI exams.

Methods:

This is a prospective, single-center, open-label, non-randomized, single-arm trial with a historical control group (1:2). In the trial group, the investigators will recruit 100 adult AIS patients presenting during working hours, who are potentially eligible for IVT and/or EVT therapies and can be treated within 6 hours of symptom onset; all workflow will be the same with standard care according to contemporary guidelines, except that patient triage procedures related to diagnosis of ischemic stroke, differentiation of intracranial hemorrhage and identification of LVO will be conducted at ESU using lfMRI. A historical control group of 200 patients managed by standard workflow (using CT brain for imaging assessment), in the 2 years before start of this study, will be drawn from our prospective IVT/EVT registry.

The investigators shall collect clinical data at baseline, 24 hours, 72 hours, 5 days, 7 days, discharge (or 14 days if earlier), and 90 days. Patients will also receive follow-up lfMRI exams at 24 hours, 72 hours, 5 days, 7 days, 14 days (or discharge). The primary outcome is DNT (min) for IVT. Main secondary outcomes include DPT (min) for EVT, proportions of patients receiving IVT and/or EVT therapies, door-to-recanalization time for EVT, mRS and NIHSS at discharge (or 14 days), mRS at 90 days, and costeffectiveness analysis. Main safety outcomes include symptomatic intracranial hemorrhage within 36 hours, before discharge (or 14 days) and within 90 days, and mortality, adverse events, severe adverse events within 90 days. Imaging outcomes include changes of infarct volume over time, and changes/emergence of hemorrhagic transformation.

Significance:

Findings from this project and subsequent efforts could help reshape and improve the efficiency of IVT/EVT patient triage at AED, which will ultimately benefit stroke patients and the stroke care system in Hong Kong and elsewhere.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years;
2. Diagnosed as ischemic stroke;
3. Potentially eligible for IVT and/or EVT and can be treated within 6 hours of symptom onset (time of symptom onset is defined as the last known normal time);
4. Presenting to AED during working hours (8AM to 6PM, weekdays);
5. Written informed consent from patients or representatives, who understand Cantonese, to participate in this study.

Exclusion Criteria:

1. Patients with unstable vital signs who need urgent medical interventions/care;
2. Confirmed contraindications for IVT or EVT by initial assessment (e.g., unstable vital signs, history of severe head trauma within 3 months, known bleeding tendency), before starting brain imaging exams;
3. Claustrophobia or other conditions that are contraindicated for MRI;
4. Patients with pacemakers, brain stimulators or insulin pumps;
5. Patients with medical or other conditions that prevent cooperation with the procedures;
6. Pregnant or breastfeeding women;
7. Participation in other clinical trials within 3 months before screening.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-12-02 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Door-to-Needle time(min) for intravenous thrombolysis | Day 0
  Reduction in the Door-to-Needle time(min) for intravenous thrombolysis

SECONDARY OUTCOMES:
Door-to-Groin Puncture time (min) for endovascular thrombectomy (EVT) | Day 0
  Reduction in the Door-to-Groin Puncture time (min) for endovascular thrombectomy
Time from symptom onset to decision for IVT/EVT (min) | Day 0
  Reduction in time from symptom onset to decision for IVT/EVT (min)
Time from admission to decision for IVT/EVT (min) | Day 0
  Reduction in time from admission to decision for IVT/EVT (min)
Improvement in NIHSS score at 24 hours compared to baseline | From Day 0, post treatment, to Day 1.
  30% improvement in NIHSS score at 24 hours compared to baseline
modified Rankin Scale (mRS) | From Day 0 post treatment, up to 90 Days.
  mRS 0-1 at discharge (or 14±2 days), and at 90±7 days ; mRS 0-2 at discharge (or 14±2 days), and at 90±7 days ; mRS distribution at discharge (or 14±2 days), and at 90±7 days
Proportion of patients receiving reperfusion therapy (including standalone IVT, standalone EVT and bridging therapy) | Day 0
  Proportion of patients receiving reperfusion therapy (including standalone IVT, standalone EVT and bridging therapy)
Door-to-reperfusion time (min) in EVT | Day 0
  Door-to-reperfusion time (min) in EVT

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Wai Hong LEUNG, MD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No